CLINICAL TRIAL: NCT06539689
Title: A Prospective, Multicenter and Randomized Controlled Trial to Evaluate the Efficacy and Safety of Sperstent® Peripheral Spot Stent System Used for the Residual Lesions After Percutaneous Transluminal Angioplasty of Femoropopliteal Arteries
Brief Title: A Trail of Sperstent® Used for Residual Lesions of Femoropopliteal Arteries
Acronym: SURF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FrontAce Scientific Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FA001
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Arterial Disease; Stenosis; Dissection
Keywords: Peripheral Arterial Disease; Spot stent
MeSH Terms: conditions — Peripheral Arterial Disease; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sperstent® peripheral spot stent system (Experimental): subjects using the Sperstent® peripheral spot stent system
  Interventions: Device: Sperstent® peripheral spot stent system
- Everflex® self-expanding peripheral stent system (Active Comparator): subjects using the Everflex® self-expanding peripheral stent system
  Interventions: Device: Everflex® self-expanding peripheral stent system

INTERVENTIONS:
Device: Sperstent® peripheral spot stent system — Sperstent® peripheral spot stent system, Percutaneous Transluminal Angioplasty (PTA), Digital Subtraction Angiography（DSA）
  Arms: Sperstent® peripheral spot stent system
Device: Everflex® self-expanding peripheral stent system — Everflex® self-expanding peripheral stent system, Percutaneous Transluminal Angioplasty (PTA), Digital Subtraction Angiography（DSA）
  Arms: Everflex® self-expanding peripheral stent system

SUMMARY:
This is a prospective, multi-center, randomized trial designed to investigate the efficacy and safety of Sperstent® peripheral spot stent system versus Everflex® self-expanding peripheral stent system in the endovascular treatment of post-balloon angioplasty (post-PTA) residual lesions including stenoses and/or dissections in femoral and proximal popliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years old, male or female;
* The target lesion is located in the superficial femoral artery or the proximal popliteal artery;
* Peripheral arterial stenosis or occlusive disease with symptoms consistent with the Rutherford classification 2 to 5;
* Estimated life expectancy >1 year;
* Subject has been informed of and understands the nature of the study and provides signed informed consent to participate in the study.

Angiographic Inclusion Criteria:

* Stenosis rate ≥70% under DSA by visual estimate, or 100% occluded lesion with a total lesion length less than 150mm (by visual estimate);
* Reference vessel diameter is between 3 mm and 7.5 mm, 50mm≤Total cumulative length of target lesions≤250mm; (In the case of bilimb lesions, a single target lesion with one limb meeting the protocol criteria is selected by the investigator; More than 2cm between lesions are considered as 2 lesions);
* After PTA treatment by DCB, there exists residual lesions, such as the target lesion has over 30% residual DS and/or presence of at least one post-PTA dissection (Type A-F) (by visual estimate);
* Patients with unobstructed inflow tract or successfully treated, visual residual stenosis ≤50%;
* Angiography showed at least one outflow tract was unobstructed at the distal end (Stenosis degree ≤70% before intervention).

Exclusion Criteria:

* Target vessel had undergone open surgery such as bypass surgery or the target lesion is in-stent restenosis;
* Patients with serum creatinine >2.5mg/dl during screening or undergoing long-term hemodialysis or peritoneal dialysis;
* Severe coagulation disorder;
* Patients with major vascular-related diseases, including acute lower extremity ischemia, active disseminated intravascular coagulation, thromboangiitis obliterans, deep vein thrombosis, and aneurysms of therapeutic lateral vessels (deep femur, superficial femur, or popliteal artery);
* A history of major organ failure or other serious illness (including severe coronary heart disease, severe cardiac insufficiency, severe neurosis, or mental illness); Have received or plan organ transplantation, severe gastrointestinal bleeding);
* Myocardial infarction or symptomatic stroke occurred within 3 months prior to enrollment;
* Thrombolysis of target vessel within 72 hours before surgery, did not completely dissolve the thrombus;
* Systemic infection or uncontrolled infection within the target limb;
* Known allergy to contrast agents, nickel or titanium (Nitinol), heparin, aspirin, clopidogrel, anesthetics;
* Women who are pregnant or breast-feeding, or women of childbearing age who have family plans within 1 year;
* Patients who are planning to have major lower limb amputations on the target side of the lesion;
* Endovascular or surgical procedures are performed on the target limb within 30 days before or 30 days after surgery;
* Participating in clinical trials of other medical devices or drugs;
* The investigator considers the patient is not suitable for participation in the clinical trial.

Angiographic Exclusion Criteria:

* Failure of the guidewire to pass through the lesion；
* During the procedure, the target lesions had received or were scheduled to receive volume reduction procedures such as cryogenic angioplasty, laser angioplasty, and percutaneous intracavity plaque gyrotomy；
* The target lesion before stent implantation is thrombotic obliteration, which is not suitable for stent implantation；
* The target lesions were severely calcified and could not fully predilate; Or grade 4 calcification；
* Acute vascular occlusion or acute or subacute thrombosis in the target lesion；
* Stent was implanted into the target vessel before enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-12-04 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Patency | 12 months post-operation
  Primary patency defined as freedom from clinically driven target lesion revascularization (CD-TLR) and freedom from duplex ultrasound derived binary restenosis at 12 months post-operation.(defined as PSVR >2.5)
Freedom from Major Adverse Events (MAEs) | 30 days post-operation
  Freedom from the occurrence of any new-onset MAEs defined as all-cause death, index limb amputation (above the ankle), or clinically-driven target lesion revascularization (CD-TLR) at 30 days post-operation.

SECONDARY OUTCOMES:
Rate of Device Success | immediately post-operation
  Defined as successful delivery, release and retrieval of the device.
Rate of Procedural Success | immediately post-operation
  Demonstrated vessel patency (<30% residual DS, by visual estimate) without the use of a bailout stent or the occurrence of MAE upon completion of the index procedure.
Primary Patency at 30 days and 6 months | 30 days and 6 months post-operation
  defined as freedom from clinically driven target lesion revascularization (CD-TLR) and freedom from duplex ultrasound derived binary restenosis at 30 days and 6 months post-operation (defined as PSVR >2.5)
Rate of clinically driven target lesion revascularization (CD-TLR) | 30 days, 6 months and 12 months post-operation
  Clinically driven target lesion revascularization (CD-TLR) was defined as an endovascular reintervention performed for a >50% diameter stenosis of the target vessel in the presence of a recurrent PAD symptom after the initial endovascular procedure.
Changes from Baseline in Rutherford Classification | 30 days, 6 months and 12 months post-operation
  Defined as change in target limb Rutherford class from baseline. Rutherford Classification is defined as follows, with increasing severity:
  Rutherford Category 0 - Asymptomatic. Rutherford Category 1 - Mild Claudication. Rutherford Category 2 - Moderate Claudication. Rutherford Category 3 - Severe Claudication. Rutherford Category 4 - Ischemic Rest Pain. Rutherford Category 5 - Minor Tissue Loss (minor exertion). Rutherford Category 6 - Major Tissue Loss (gangrene).
Changes from Baseline in Ankle-brachial Index (ABI) | 30 days, 6 months and 12 months post-operation
  Defined as change of target limb ABI from baseline. The Ankle Brachial Index (ABI) is the systolic pressure at the ankle, divided by the systolic pressure at the arm.
Duplex Ultrasound (DUS) Derived Lesion Patency | 30 days, 6 months and 12 months post-operation
  Lesion Patency is evaluated by Duplex Ultrasound (DUS)
Rate of major adverse event(s) (MAEs) | 6 months and 12 months post-operation
  MAEs defined as all-cause death, index limb amputation (above the ankle), or clinically-driven target lesion revascularization (CD-TLR) .
Rate of Stent Fracture | 12 months post-operation
  Stent fractures will be analyzed by X-ray at 12 months post-operation. The stents implanted into a certain subject will be analyzed collectively in the assessment. Stent fractures will be assessed with Grade I, II, III or IV as follow.
  Grade I - a single strut fracture only. Grade II - multiple single strut fractures that occur at different sites of a stent or different stents.
  Grade III - multiple nitinol stent fractures resulting in complete transverse linear fracture.
  Grade IV - a spiral dissection of a stent. Fractures of Grade I are least severe, increasing in severity to Grade IV.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Liyuan Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Hospital of Chengdu University of TCM, Chengdu
  - Shanghai East Hospital, Shanghai